CLINICAL TRIAL: NCT06447935
Title: Acute Eosinophilic Myocarditis International Registry
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NIGUARDA H
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Myocarditis
Keywords: Eosinophilic Myocarditis; Endomyocardial Biopsy
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Eosinophilic Myocarditis: Patients affected by Acute Eosinophilic Myocarditis with the following inclusion criteria:
  1. histologically EM proven "borderline" (presence of inflammatory infiltrate) or "active" (presence of inflammatory infiltrate plus myocardial necrosis) myocarditis, according to the Dallas criteria;
  2. acute presentation defined by the onset of cardiac symptoms within 30 days before admission.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — not applicable - no intervention required

SUMMARY:
Retrospective collection of clinical, histological, imaging data regarding patients with acute histologically-proven eosinophilic myocarditis.

DETAILED DESCRIPTION:
Eosinophilic myocarditis (EM) is an acute life-threatening inflammatory disease of the heart. We collect clinical, histologic, laboratory, diagnostic and imaging data regarding acute EM with a histological diagnosis and symptoms onset within 30 days from first medical contact from hospitals around the world. The main objective is to investigate and describe clinical presentation, main systemic conditions associated and outcomes of the first series of patients with acute myocarditis and histological evidence of eosinophilic infiltration within myocardium.

ELIGIBILITY:
Patients with histological diagnosis gained during an hospitalization within 30 days from symptoms onset.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective observational cohort of eosinophilic myocarditis patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Natural History of Eosinophilic Myocarditis | 3 year
  Proportion of patients who die or need a heart transplantation from index admission.

SECONDARY OUTCOMES:
Natural History of Eosinophilic Myocarditis subgroups based on etiology | 3 years
  Proportion of patients who die or need a heart transplantation from index admission dividing patients based on the underlying condition (for instance idiopathic, hypersensitivity, eosinophilic granulomatosis with polyangiitis,…)

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ammirati E, Palazzini M, Lehtonen J, Potena L, Mayranpaa MI, Ragback J, Foa A, Uribarri A, Thiele H, Vidal-Burdeus M, Freund A, Gustafsson F, Tschope C, Elsanhoury A, Ihle J, Rudi WS, Grabmaier U, Merlo M, Melenovsky V, Weislova I, Jellinghaus S, Linke A, Baldovini C, Adorisio R, Kuchynka P, Palecek T, Krejci J, Poloczkova H, Caterino AL, Gilotra NA, Lovell JP, Macomb EP, Shih J, Hong K, Rossi VA, Ruschitzka F, Cavallini C, Riccini C, Kamal M, Huang F, Groh M, Gentile P, Garascia A, Lala A, Shimokawa H, Vandenbriele C, Sionis A, Schmidt M, Grosu A, Bollano E, Turco A, Crespo-Leiro MG, Couto-Mallon D, Cannata A, Bromage DI, Narducci ML, Cicchitti V, Ianni U, De Luca L, Mistrulli R, Frea S, Raineri C, Schroeder JW, Arias AM, Emdin M, Corda M, Pasqualucci D, Greulich S, Gawaz M, Manuylova T, Martinez-Selles M, Hernandez Perez FJ, Martin Centellas A, Dominguez F, Gaillet A, D'Alessandris N, Trankle C, Halushka MK, Moroni F, Abbate A, Basso C, Sinagra G, Veronese G, Camici PG, Adler ED, Bernasconi DP, Klingel K, Cooper LT Jr. Natural History of Patients With Histologically Proven Acute Eosinophilic Myocarditis. Circulation. 2026 Feb 6. doi: 10.1161/CIRCULATIONAHA.125.074797. Online ahead of print. PMID 41645905